CLINICAL TRIAL: NCT01820234
Title: Evaluation of Store-and-Forward Teledermatology Versus a Face-to-Face Assessment During a Skin Cancer Screening Event
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 201018315
Record Dates: First submitted 2011-02-04; First posted 2013-03-28 (Estimated); Last update posted 2017-07-19 (Actual); Status verified 2013-03

CONDITIONS: Skin Cancer; Screening; Telemedicine
Keywords: Skin cancer; Teledermatology; Screening; Store-and-forward
MeSH Terms: conditions — Skin Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- In-person dermatology evaluation (Other): Health care modality
  Interventions: Other: In-person dermatology evaluation
- Store-and-forward teledermatology evaluation (Other): Health care modality
  Interventions: Other: Store-and-forward teledermatology evaluation

INTERVENTIONS:
Other: In-person dermatology evaluation — Every patient will be evaluated by an in person dermatologist present at the screening.
  Arms: In-person dermatology evaluation
Other: Store-and-forward teledermatology evaluation — Every patient will be evaluated online via a store and forward teledermatology modality.
  Other Names: Health care modality
  Arms: Store-and-forward teledermatology evaluation

SUMMARY:
The purpose of this study is to determine the diagnostic and management concordance of face-to-face dermatologist versus a store-and-forward teledermatologist at a skin cancer screening event.

The investigators' hypotheses include the following:

1. Compared to in-person assessment, store-and-forward teledermatology assessment will result in adequate diagnostic concordance.
2. Compared to in-person assessment, store-and-forward teledermatology results in adequate management concordance.
3. The sensitivity and specificity of store-and-forward evaluation to detecting lesions that are either premalignant or malignant will be similar to that of in-person evaluation.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older at time of consent, may be male or female.
* Able to provide a brief medical history and have/allow an examination of their skin including photographs.
* Capable of giving informed consent.
* Will be able to receive notification of follow-up recommendations

Exclusion Criteria:

* Patients who will not provide informed consent
* Patient who are unable to fulfill tasks of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2010-09; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Aggregated diagnostic concordance | At the time of dermatologist evaluation (Day 1)
  Aggregated diagnostic concordance which is defined as the agreement of the in-person dermatologist's principle diagnosis with the teledermatologist's primary diagnosis or any of the differential diagnoses.

SECONDARY OUTCOMES:
Primary diagnostic concordance | At the time of dermatologist evaluation (Day 1)
  Diagnostic concordance between the in-person dermatologist and the teledermatologist for their primary diagnosis.
Categorical diagnostic concordance | At the time of dermatologist evaluation (Day 1)
  Diagnostic concordance between the in-person dermatologist and teledermatologist based on standard clinical diagnostic categories for each lesion.
Management concordance | At the time of dermatologist evaluation (Day 1)
  The concordance between the in-person dermatologist and teledermatologist for the chosen management plan for each lesion.
Sensitivity | At the time of dermatologist evaluation (Day 1)
  The sensitivity of store-and-forward evaluation to detecting lesions that are either premalignant or malignant.
Specificity | At the time of dermatologist evaluation (Day 1)
  The specificity of store-and-forward evaluation to detecting lesions that are either premalignant or malignant.

CONTACTS AND LOCATIONS:
Overall Officials: April W Armstrong, MD, MPH, Principal Investigator — University of California, Davis
Locations (1):
- University of California, Davis Shifa Community Clinic, Sacramento, California, United States